CLINICAL TRIAL: NCT00386815
Title: Safety Confirmation Study of LY231514 Plus Cisplatin in Patients With Malignant Pleural Mesothelioma
Brief Title: Safety Confirmation Study of Pemetrexed Plus Cisplatin in Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10512; H3E-JE-ME02
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Malignant Pleural Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Pemetrexed; Cisplatin

INTERVENTIONS:
Drug: pemetrexed
Drug: cisplatin

SUMMARY:
To investigate safety of pemetrexed combined with cisplatin for chemo therapy-naive patients with malignant pleural mesothelioma

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of malignant pleural mesothelioma
* Not candidates for curative surgery. Patients will be clinically staged using the IMIG TNM staging criteria
* Not receive prior systemic chemotherapy
* Patients must have measurable lesions, which are diagnosed by CT, or MRI scan within 28 days before administration
* More than 20 years and less than 75 years of age
* ECOG Performance status score: 0 - 1
* Prior radiation therapy is allowed to < 25% of the bone marrow. Prior radiotherapy must be completed at least 21 days before study enrollment, and the patients must have recovered from the toxic effects of the treatment prior to study enrollment.
* Prior surgeries must be completed at least 21 days before study enrollment, and the patients must have recovered from the effects of the operation.However, regarding examination of thoracotomy or celiotomy, etc. if the investigator or sub-investigator judges that there are no influences of surgery and no problems for participation of patients in this study, e.g. safety security, there should be at least 14 days from the surgery day to patient registration date
* Patients who have adequate organ function Hemoglobin: no less than 9g/dl, Absolute neutrophil count: no less than 2,000/mm3, Platelet count: no less than 100,000/mm3,Serum albumin: no less than 2.5g/dL,AST (GOT) and ALT (GPT): no more than 2.5 x the upper limit of reference values at each site (no more than 5 x the upper limit of reference values at each site is acceptable if liver has tumor involvement), Total bilirubin: no more than 1.5 x the upper limit of reference values at each site,Serum creatinine: no more than the upper limit of reference values at each site, SpO2: no less than 92%, ECG: normal (In the case of the ECG was marked abnormal waveshape, when the investigator or sub-investigator judges that there is no safety issue for the patient, administration can be done), 24hr-creatinine clearance or calculated creatinine clearance: no less than 45mL/min
* Estimated life expectancy of at least 90 days from the registration date
* Patients must be hospitalized from the start of the first cycle until the start of the second cycle of the combination therapy, in principle (Only in case investigator or sub-investigator judges that there are no safety issues, patients can receive the therapy as outpatients from the middle of Cycle 1)
* Male and female patients with reproductive potential must use an approved contraceptive method if appropriate (eg, intrauterine device [IUD], birth control pills, or barrier device) during and for 90 days after study therapy. Females with childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to study enrollment.
* Signed informed consent from patient

Exclusion Criteria:

* Serious or uncontrolled concomitant systemic disorders
* Active systemic infection
* Active, double cancer (patients with synchronous double cancers or asynchronous double cancers with non-disease period of no more than 5 years)(except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Patients who have symptomatic brain metastases or those who have brain metastases which require treatment
* Presence of clinically detectable third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Having a history of sensitivity to platinum agent, folic acid or vitamin B12
* Women who are pregnant, breast-feeding or could be pregnant or women who hope to get pregnant during or within 90 days after the study.
* Man who hopes their partner will become pregnant during or within 90 days after the study.
* Patients who have neurotoxicity which is no less than CTC grade 2 at study entry.
* Inability to interrupt salicylates of other nonsteroidal anti-inflammatory agents for a 5-day period(8-day period for long-acting agents such as piroxicam).
* Inability and unwillingness to take folic acid or vitamin B12 supplementation.
* Plane chest X-rays show widely diffuse images that have been caused by interstitial pneumonia.
* Patients who have been judged inadequate for the study by the investigator or sub-investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To investigate safety profile when administered pemetrexed combined with cisplatin in malignant pleural mesothelioma patients

SECONDARY OUTCOMES:
To investigate efficacy when administered pemetrexed combined with cisplatin in malignant pleural mesothelioma patients

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- Japan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com